CLINICAL TRIAL: NCT06239922
Title: Establishing Cognitive and Neural Assessment Platform and Localized Norm for Macau Older Adults
Brief Title: Cognitive and Neural Assessment Platform and Localized Norm for Macau Older Adults.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Macau (Other)
Responsible Party: Sponsor
Other Study IDs: BSERE23-APP019-ICI; 0153/2022/A (Other Grant/Funding Number: The Science and Technology Development Fund (FDCT)of the Macao Special Administrative Region (SAR))
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Cognition Disorders in Old Age; Cognitive Decline; Cognitive Impairment; Cognitive Dysfunction; Cognitive Change; Aging
Keywords: Macau; cognitive aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Older adults
- Group 2: Younger adults

SUMMARY:
The current project is dedicated to creating a comprehensive cognitive and neural assessment platform and corresponding norms tailored specifically to the older adults in Macau.

DETAILED DESCRIPTION:
The investigators will establish this assessment platform using a combination of methods, including interviews, surveys, and expert reviews.

Steps include adapting existing assessment methods to the Macau context, developing new cognitive and neural tasks, defining standardized procedures, seeking external expert input, conducting pilot tests, and validation processes, and refining both the platform and its accompanying manual.

ELIGIBILITY:
Inclusion Criteria:

* Must be a local adult resident of Macau
* Age above 50 years for older adult cohort
* Younger adults individuals above 18 will be included as control comparators

Exclusion Criteria:

* History of neurological injury or disease
* Current use of medications that affect brain function or blood flow
* Contraindications to MRI scanning, such as the presence of an electric/mechanical implant or device (e.g., pacemaker)
* Claustrophobia
* Body weight over 300 lbs due to weight and physical constraints of the scanner (i.e., bore size limited to 55 cm)
* Inability to provide informed consent
* Pregnancy
* Being under the legal age of adulthood (children)
* Incarcerated individuals (prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults above 50 years old from the Macau local community.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Normative Data for the Montreal Cognitive Assessment - Chinese (Hong Kong) version | From February 2024 to January 2026
  The MoCA will be administered to derive a normative data set representative of the older adult population in Macau.
Normative Data for the Mini-Mental State Examination (MMSE) | From February 2024 to January 2026
  The MMSE will be administered to derive a normative data set representative of the older adult population in Macau.
Normative Scores for Computerized Neuropsychological Tasks | From February 2024 to January 2026
  Neuropsychological tasks will be employed to measure selective attention capacity and processing speed in the study cohort. These tasks will provide quantifiable data on the efficiency and accuracy of cognitive processing. The collective performance on these tasks will be used to establish benchmark values - including means, medians, and ranges - that define the normative standards for these cognitive abilities in the population.

SECONDARY OUTCOMES:
Neural Activation Patterns During Cognitive Tasks as Revealed by Functional Magnetic Resonance Imaging (fMRI) | From February 2024 to January 2026
  fMRI data will be collected to identify patterns of neural activation associated with cognitive task performance.
Cerebral Hemodynamics Assessed Through Functional Near-Infrared Spectroscopy (fNIRS) | From February 2024 to January 2026
  fNIRS will be employed to measure cerebral blood flow and oxygenation during cognitive tasks.
Electrophysiological Correlates of Cognitive Activity as Measured by Electroencephalography (EEG) | From February 2024 to January 2026
  EEG will be utilized to record the electrical activity of the brain during cognitive tasks. Key outcome metrics will include event-related potentials (ERPs) amplitudes and latencies, with mean values and variability measures reported for the cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Haoyun ZHANG Assistant Professor, Ph.D, Principal Investigator — University of Macau
Locations (1):
- Centre for Cognitive and Brain Sciences of the University of Macau, Macao, Macao SAR, Macau

IPD SHARING:
Plan to Share IPD: Undecided